CLINICAL TRIAL: NCT06245070
Title: Immediate and Short-term Effects of High-definition Transcranial Direct Current Stimulation Over the Left Supplementary Motor Area on Voice and Speech Functions in Parkinson's Disease
Brief Title: Speech and Voice Outcomes Following HD-tDCS Over the Left SMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRBAM-21-1019
Record Dates: First submitted 2024-01-24; First posted 2024-02-07 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Brain stimulation; Supplementary motor area; Speech; Voice
MeSH Terms: conditions — Parkinson Disease; Speech

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active high definition transcranial direct current stimulation (HD-tDCS) (Experimental): High-definition anodal transcranial direct current stimulation (2 milliamps [mA]) for 5 consecutive days (one session per day for 20 minutes each). The electrical current will be administered over the left Supplementary motor area. The stimulation will be delivered at an intensity of 2 milliamps (mA) for a maximum of 20 minutes.
  Interventions: Device: Active transcranial direct current stimulation
- Sham high definition transcranial direct current stimulation (HD-tDCS) (Experimental): High-definition sham transcranial direct current stimulation (2 milliamps [mA]) for 5 consecutive days (one session per day for 20 minutes each). The electrical current will be administered over the left Supplementary motor area. The current will be ramped up for the first 30 seconds following which the intensity will drop to 0 milliamps (mA).
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Active transcranial direct current stimulation — HD electrodes (diameter of 1.2 cm) will be placed on the participants' skull using an HD-tDCS cap (Soterix Medical Inc. New York) and based on 5-10 international montage. Active stimulations will be delivered by a 9 MxN Soterix HD-tES device for 20 minutes( 2 mA) per day for 5 days.
  Arms: Active high definition transcranial direct current stimulation (HD-tDCS)
Device: Sham transcranial direct current stimulation — HD electrodes (diameter of 1.2 cm) will be placed on the participants' skull using an HD-tDCS cap (Soterix Medical Inc. New York) and based on 5-10 international montage. Sham stimulations will be delivered by a 9 MxN Soterix HD-tES device. In the sham tDCS condition, the current is only on for 30 seconds before it is ramped back down to 0 milliamps (mA), although the electrodes are still worn for 20 minutes.
  Arms: Sham high definition transcranial direct current stimulation (HD-tDCS)

SUMMARY:
Pharmaceutical and neurosurgical treatments reliably ameliorate the cardinal motor symptoms in PD but, they often yield inconsistent outcomes for speech and voice disorders, with some studies showing exacerbation of pre-treatment deficits. Therefore, it is crucial to develop and optimize novel approaches that could simultaneously improve speech and voice deficits in PD and facilitate existing behavioral interventions. This project will investigate the immediate and short-term effects of multiple sessions of HD-tDCS over the left SMA on speech and voice deficits in PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a movement disorder that affects more than one million individuals in the United States. Over 90 percent of individuals with PD manifest speech and voice impairments in the course of their disease, which can significantly compromise patients' quality of life. While pharmaceutical intervention and deep brain stimulation reliably improve the cardinal motor symptoms of PD, such as tremor, rigidity, and bradykinesia, the effects of these treatments on speech and voice are inconsistent, with some studies showing the exacerbation of pre-treatment deficits. This inconsistency often occurs because treatments are calibrated to ameliorate limb motor symptoms, with no direct optimization to improve speech and voice functions. However, there is no established non-invasive neurostimulation protocol for communication disorders in PD. Increasing evidence supports the application of non-invasive brain stimulation techniques such as transcranial direct current stimulation (tDCS) to improve both motor and non-motor symptoms in PD. However, limited evidence exists regarding the application of tDCS to improve speech and voice disorders in PD. Moreover, there is no established long-term effect of tDCS on speech and voice deficits in PD. In this proposed study, we will address these gaps by investigating the immediate and short-term effects of high definition-transcranial direct current stimulation (HD-tDCS) over the left supplementary motor area (SMA) on speech and voice deficits in 24 PD and 24 matched control participants.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Native English speakers
* Adequate age-relative hearing and vision to perform the outlined tasks
* Able to provide their own written consent

Exclusion Criteria :

* Neurological disorders besides Parkinson's disease
* Previous brain surgery including deep brain stimulation
* Clinical diagnosis of dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-02 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Voice loudness measures | Acoustic measures related to voice loudness will be measured at baseline, immediately after the last session of stimulation, one week and one month after the las stimulation session.
  Acoustics measures of voice loudness including voice intensity (dB), shimmer (Cycle-to-cycle voice intensity perturbation) and smoothed cepstral peak prominence will be calculated for each participant.
Fundamental frequency measures | Fundamental frequency (F0), jitter (Cycle-to-cycle voice F0 perturbation) and harmonic to noise ration will be calculated for each participant.
  Changes in the accuracy rate (percentage of correct repetitions) of non-word repetition
Accuracy of syllable repetition | Accuracy rate for syllable repetition will be measured at baseline, immediately after the last session of stimulation, one week and one month after the las stimulation session.
  The number of syllables that correctly produced during syllable repetition task will be calculated for each participant.
Speech rate | Speech rate will be measured at baseline, immediately after the last session of stimulation, one week and one month after the las stimulation session.
  The speech rate ( number of syllables per second) will be calculated during a syllable repetition task for each participant.
Speech rate stability | Speech rate stability will be measured at baseline, immediately after the last session of stimulation, one week and one month after the las stimulation session.
  Variability in speech rate across trials for each syllable length ( 1, 2, and 3 ) will be calculated for each participant.

IPD SHARING:
Plan to Share IPD: No
Participants' data are confidential. de-identified data will be publicly available after final analysis.